CLINICAL TRIAL: NCT02484209
Title: A 16 Week PILOT Study to Determine the Frequency of Sulphonylurea-Associated Hypoglycaemia in Older Moderately Frail Patients With Type 2 Diabetes Mellitus Poorly Controlled on Metformin: an Open Label Study ( DIAFRAIL Study)
Brief Title: DiaFrail: A Short Duration Study in Older People ( DIAFRAIL Study)
Acronym: DiaFrail
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Inclusion criteria too strict making it difficult to recruit in primary care
Sponsor: Diabetes Frail Ltd (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Caroline Sinclair, Professor Alan Sinclair - Principal Investigator, Director of Diabetes Frail Ltd, Diabetes Frail Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DF-07
Record Dates: First submitted 2015-06-15; First posted 2015-06-29 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; frailty; aged; metformin; sulphonylurea; hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus; Frailty; Hypoglycemia | interventions — Metformin; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride + metformin (Experimental): Glimepiride (2-4mg twice daily) + metformin (1500 mg daily) (n = 10 in total) Older subjects with moderate frailty will be assigned for 16 weeks to this arm. A subgroup (n=5) will undergo 3 x 72h periods of CBGM
  Interventions: Drug: Glimepiride; Drug: Metformin
- Metformin (Active Comparator): Metformin (1500 mg daily) (n = 10 in total) Older subjects with moderate frailty will be assigned for 16 weeks to this arm. A subgroup (n=5) will undergo 3 x 72h periods of CBGM
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 1500 mg daily for 16 weeks
  Other Names: glucophage
  Arms: Metformin
Drug: Glimepiride — glimepiride 2-4 mg twice daily for 16 weeks
  Other Names: Amaryl
  Arms: Glimepiride + metformin
Drug: Metformin — metformin 1500 mg daily for 16 weeks
  Other Names: Glucophage
  Arms: Glimepiride + metformin

SUMMARY:
1. Many patients with type 2 diabetes are not at glycaemic goal and require additional therapy in order to reduce vascular risk and improve symptom control
2. Sulphonylurea therapy is a commonly prescribed 2nd-line glucose -lowering agent and its use is recommended in major clinical guidelines for diabetes and also in the recently presented IDF (International Diabetes Federation) guidelines for older people.
3. Older people with diabetes are not a homogeneous group and as many as 25% are frail.
4. Frailty is a PRE-DISABILITY state but may increase the 'vulnerability' of many older people to having a fall, admission into hospital, or perhaps increasing their risk of hypoglycaemia
5. As a consequence of their glucose-lowering ability, sulphonylureas may increase the risk of hypoglycaemia in older people and those who have features of frailty may be at increased risk.
6. The investigators therefore need to estimate the risk of hypoglycaemia in moderately frail older subjects with type 2 diabetes who are taking sulphonylurea therapy as this is a commonly prescribed class of agent used routinely in clinical practice
7. Thus, this short term project wishes to assess the frequency of hypoglycaemia in subjects with some evidence of frailty with type 2 diabetes by a series of glucose monitoring techniques with excellent research team support to minimize any safety issues. An identical study at the Second University of Naples, Italy under the supervision of Professor Giuseppe Paolisso is planned and is the second study site for this PILOT project.

DETAILED DESCRIPTION:
Rationale for Study

The rates of hypoglycaemia in older people with diabetes are not known with any accuracy and there are no data in older frail patients with diabetes. However, as this latter group is increasingly recognized as a specific subgroup of patients with diabetes it is important to assess how safe sulphonylurea agents are in older patients as this group of glucose-lowering medication is recommended in most diabetes clinical guidelines including algorithms.

The data for rates of mild to moderate hypoglycemia in older people with diabetes is also very scant and because many episodes may be asymptomatic, these take place without either the patient or family knowing, and thus important information of this nature does not reach the clinician in charge of prescribing. In these latter circumstances, continuous blood glucose monitoring (CBGM) will have an important role to detect the frequency of these episodes and will be used in a subgroup of each treatment arm in this PILOT study. When hypoglycaemic episodes are accompanied with symptoms, detection rates are obviously improved. It is important note that even mild symptomatic hypoglycemia may be associated with increased cardiovascular events, increased hospitalisation and increased mortality although this study was in a young 'elderly' group (average age about 63y), There is thus an important need to assess what this risk is and whether commonly used sulphonylureas are relatively safe in this respect. As metformin and sulphonylureas are still the commonest agents used to lower glucose levels in people with diabetes, the investigators wish to study these first in our programme of studies in this area. With the development of other classes of oral glucose-lowering agents such as DPP4-inhibitors which are associated with low levels of hypoglycaemia and are well tolerated in older patients with type 2 diabetes (5), it is important to provide more justification for their use by discovering if hypoglycaemia, both subclinical/asymptomatic and more serious forms of hypoglycaemia occur commonly in sulphonylurea treatment.

The data for rates of mild to moderate hypoglycemia in older people with diabetes is even more scant - when symptomatic, detection rates are improved, but when asymptomatic, detection requires CBGM. In a young 'elderly' group (average age about 63y), even mild symptomatic hypoglycemia may be associated with increased cardiovascular events, increased hospitalisation and increased mortality Therefore, the primary object of this short PILOT hypoglycemia rate-determining study will be the evaluation of the difference (as % of variation of mild-moderate hypoglycemic events) between glimepiride (2-4mg twice daily) as add on to metformin, and metformin treatment alone (at maximal dose (1500 mg/day), in mild to moderately frail older type 2 diabetic patients aged over 70 years. The investigators will wish to observe whether the intervention group has had a change in HbA1c levels during the treatment period with glimepiride.

ELIGIBILITY:
Inclusion Criteria:

1. Frail older patients with type 2 diabetes without adequate glycemic control (HbA1c >8.0%, >64 mmol/mol) while on metformin treatment. A previous diagnosis of type 2 diabetes mellitus will have met ADA criteria. Frailty will be identified by using the easy to use Clinical Frailty Scale (see appendix) with patients being described as point 4 (vulnerable), or point 5 (mildly frail), or point 6 (moderately frail (18).
2. Patient understands the study procedures, alternative treatments available, and risks involved with the study, and voluntarily agrees to participate by giving written informed consent.
3. Patient is a male or female and >70 years of age on the day of signing informed consent.

Exclusion Criteria:

1. BMI >32 Kg/m2.
2. Patient has hypersensitivity or intolerance to glimepiride or any component of this medication.
3. Patient treated with insulin.
4. Patient with severe evidence of frailty (Clinical Frailty Scale -point 7-9)
5. Patient (or carer) unable to manage SBGM (self blood glucose monitoring) and/or CBGM
6. Patient routinely consumes more than 2 alcoholic drinks per day.
7. Patient is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent.
8. Patient's glycaemia are >300 mg/dL (>16.7 mmol/l) at Visit 2.
9. Patient has uncontrolled endocrine or metabolic disease known to influence glycaemia (i.e., secondary causes of hyperglycaemia).
10. Patient has a history or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the patient's participation for the full duration of the study, such that it is not in the best interest of the patient to participate.
11. Patients with an established diagnosis of dementia
12. Patients with a memory disorder, those needing an interpreter, or those with severe visual impairment (unable to complete the tests)
13. Patient has congestive heart failure defined by NYHA (New York Heart Association) Class III or IV.
14. Patient has unstable angina pectoris.
15. Patient has had a myocardial infarction, coronary artery bypass surgery. Angioplasty or uncontrolled or severe peripheral artery disease within previous 6 months
16. Patient has had a partial ileal bypass gastric bypass, or other significant intestinal malabsorption.
17. Patient has uncontrolled hypertension (treated or untreated) with systolic blood pressure >180 mm Hg or diastolic >100 mm Hg at Visit 1. Investigators are encouraged to maximize blood pressure control according to current guidelines prior to randomization.
18. Patient has estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2 based on the 4-variable MDRD (Modification of Diet in Renal Disease) equation, nephrotic syndrome or other clinically significant renal disease at baseline..
19. Patient has a history of malignancy < 5 years prior to signing informed consent.
20. Patient is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
21. Patient has a history major psychiatric illness not adequately controlled and stable on pharmacotherapy.

    -

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2016-10 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Difference in hypoglycaemia occurrence (mild-moderate category) between treatment arms | 16 weeks
  The primary objective of this short PILOT study will be the evaluation of the difference (as % of variation of mild-moderate hypoglycaemic events) between the treatment arms

SECONDARY OUTCOMES:
Duration of Hypoglycaemia | week 1
  Duration in minutes with glucose less <54 mg/dl (3 mmol/l) during a 24-h period
Duration of Hypoglycaemia | week 8
  Duration in minutes with glucose less <54 mg/dl (3 mmol/l) during a 24-h period
Duration of Hypoglycaemia | week 16
  Duration in minutes with glucose less <54 mg/dl (3 mmol/l) during a 24-h period

CONTACTS AND LOCATIONS:
Overall Officials: Alan Sinclair, Principal Investigator — Diabetes Frail Ltd